CLINICAL TRIAL: NCT06990152
Title: Trial Clinico Randomizzato e Doppio-cieco Sull'Efficacia di Una Formulazione Alimentare Contenente Trigliceridi a Media Catena (MCT) e Fibre in Pazienti Con Artrite Psoriasica
Brief Title: A Randomized, Double-blind Clinical Trial on the Efficacy of a Dietary Formulation Containing Medium-chain Triglycerides (MCT) and Fiber in Patients With Psoriatic Arthritis
Acronym: CALIPSO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Schär AG / SPA (Industry)
Collaborators: ASST Gaetano Pini-CTO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CALIPSO-2025
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Psoriatic Arthritis (PsA)
Keywords: medium-chain triglycerides; dietary fiber; psoriatic arthritis; CALIPSO
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control placebo group (Placebo Comparator): Patients assigned to this group will consume a placebo powder.
  Interventions: Other: Placebo powder
- MCTs and fiber group (Test group) (Experimental): Patients assigned to this group will consume twice per day a portion of MCTs and fiber.
  Interventions: Other: MCTs and fiber

INTERVENTIONS:
Other: MCTs and fiber — Water-soluble powder containing medium-chain triglycerides, soluble and unsoluble fiber.
  Arms: MCTs and fiber group (Test group)
Other: Placebo powder — Water-soluble powder containing no medium-chain triglycerides and no fiber.
  Arms: Control placebo group

SUMMARY:
The primary objective of this study is to evaluate the effects of a formulation containing medium-chain triglycerides (MCTs) and vegetable fibers on the quality of life of patients with psoriatic arthritis, by monitoring the patients over a period of 3 months in a single-center interventional study. As secondary objectives, the study will assess the effects of the same formulation on disease activity and on certain blood parameters and dietary habits.

DETAILED DESCRIPTION:
The diagnostic and therapeutic framework in the field of psoriatic arthritis (PsA) is complex and not yet fully defined. Despite significant advances in pharmacological therapy and although particularly satisfactory results can be achieved thanks to new-generation DMARDs (disease-modifying antirheumatic drugs), there is still a significant gap regarding factors that, in addition to pharmacological therapy, could help patients further improve their health status, primarily dietary habits.

The aim of this study is to evaluate the effectiveness of a special medical food based on MCTs and fiber in improving quantitative and qualitative parameters in patients with PsA under stable pharmacological treatment and with low disease activity. Specifically, this will be achieved through the analysis of health-related quality of life as perceived by patients, the impact of the disease on general life, body composition and sarcopenia, physical and mental health status of patients, dietary habits, and through an evaluation of metabolic and inflammatory blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients: aged 18-80 years;
* Clinical diagnosis of PsA meeting the CASPAR classification criteria;
* Low disease activity (4 < DAPSA ≤ 14) at the time of recruitment;
* Under stable pharmacological treatment with disease-modifying antirheumatic drugs (DMARDs) (conventional synthetic, targeted synthetic, or biological);
* Disease duration > 6 months;
* Absence of metabolic diseases.

Exclusion Criteria:

* BMI ≥ 27 kg/m²;
* Current or desired pregnancies (confirmed by pregnancy test);
* Disease activity in remission (DAPSA ≤ 4), moderate (14 < DAPSA ≤ 28), or high (DAPSA > 28) at the time of recruitment;
* Pediatric onset of the disease (< 16 years);
* Patients on a vegan, ketogenic, or MCT-rich diet (containing MCT in supplement form or high amounts of palm or coconut oil);
* Presence of ketoacidosis/metabolic acidosis, decompensated liver cirrhosis, or medium-chain acyl-CoA dehydrogenase (MCAD) deficiency;
* Type 2 diabetes, cardiovascular diseases, hypertension, ischemic diseases, renal failure, malignant tumors, respiratory diseases, dyslipidemia, fibromyalgia, metabolic syndrome;
* Major depression;
* Gastritis, esophagitis, reflux syndrome, chronic inflammatory bowel diseases (IBD);
* Lactose intolerance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | baseline (T0), month 1 (T1), month 2 (T2) and month 3 (T3)
  Improvement in the health-related quality of life as perceived by patients (measured using the EuroQol-5 Dimensions-5 Levels, EQ-5D-5L, questionnaire) from baseline (T0) to the end of the study (T2) in the Test group compared to the Control group.
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (1), slight problems, moderate problems, severe problems and extreme problems (5).
  The EQ-5D-5L Index Score is derived from the descriptive system using country-specific value sets. These scores typically range from <0 (worse than death) to 1 (full health). For example, in many value sets, the minimum score can be around -0.59, and the maximum score is 1.00.
  The EQ VAS score ranges from 0 to 100, as self-reported by the patient.

SECONDARY OUTCOMES:
Impact of the disease on patient's life | baseline (T0), month 1 (T1), month 2 (T2) and month 3 (T3)
  Improvement in the impact of the disease on the patient's general life (measured using the Psoriatic Arthritis Impact of Disease 12-item questionnaire, PSAID-12) from baseline to T2 in the Test group compared to the Control group. The questionnaire includes 12 items, each representing a different domain affected by PsA, such as:
  * Pain
  * Fatigue
  * Skin problems
  * Work/leisure activities
  * Functional capacity
  * Discomfort
  * Sleep disturbance
  * Coping
  * Anxiety
  * Depression
  * Social participation
  * Overall well-being Each item is scored on a Numerical Rating Scale (NRS) from 0 to 10, where 0 means no impact and 10 indicates the highest possible impact. The total PsAID-12 score is a weighted average of the 12 items, with different weights assigned to each domain based on patient input. The final score ranges from 0 to 10, where 0 = no impact of disease and 10 = maximum impact of disease.
  Lower scores indicate better health status and lower disease impact.
Physical and mental health status | baseline (T0), month 1 (T1) and month 2 (T2)
  Changes in physical and mental health status (measured using Health Assessment Questionnaires, HAQ) from baseline to T2 in the Test group compared to the Control group.
  The Health Assessment Questionnaire Disability Index (HAQ-DI) is a widely used tool to assess functional ability in patients with rheumatic diseases, especially rheumatoid arthritis and psoriatic arthritis.
  The questionnaire includes 8 domains of daily living activities:
  * Dressing and grooming
  * Arising
  * Eating
  * Walking
  * Hygiene
  * Reach
  * Grip
  * Common daily activities Each domain contains 2-3 questions, and patients rate their difficulty performing each activity on a scale from 0 (no difficulty) to 3 (unable to do).
  If a patient uses an assistive device or needs help from another person, the minimum score for that domain is 2, unless the score is already 2 or higher.
  For each domain, the highest score among the questions is taken as the domain score. The HAQ-DI score is the average of the 8 domain scores.
Lipid profile | baseline (T0), month 1 (T1) and month 2 (T2)
  Changes in the lipid profile of patients (in terms of cholesterol, LDL, HDL, triglycerides) between T-1 and T2 in the Test group compared to the Control group.
Dietary habits | baseline (T0), month 1 (T1) and month 2 (T2)
  Changes in patients' dietary habits (assessed using the Food Frequency Questionnaire Osservatorio Grana Padano) from baseline to T2 in the Test group compared to the Control group.
Bioelectrical Impedance Analysis (BIA) | baseline (T0), month 1 (T1) and month 2 (T2)
  Changes in body composition from baseline to T2 in the Test group compared to the Control group.
  Bioelectrical Impedance Analysis (BIA) will be used to measure changes in body composition. BIA is a non-invasive, quick, and widely used method to estimate body composition, particularly:
  * Body Fat Percentage: A decrease suggests fat loss, which is often a goal in weight management or fitness.
  * Muscle Mass: An increase indicates improved strength and metabolism.
  * Visceral Fat: Lower levels reduce the risk of metabolic diseases.
  * Total Body Water (TBW): Stable or increase indicates good hydration and muscle mass.
  * Basal Metabolic Rate (BMR): An increase suggests more lean mass, which burns more calories at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Ingegnoli, Professor, Principal Investigator — ASST Gaetano Pini CTO, UOC Clinica Reumatologica
Locations (1):
- ASST Gaetano Pini CTO, UOC Clinica Reumatologica, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No